CLINICAL TRIAL: NCT00529945
Title: The Paradigm IV Trial - PFx Closure System in Subjects With Cryptogenic Stroke, Transient Ischemic Attack, Migraine or Decompression Illness
Brief Title: PFx Closure System in Subjects With Cryptogenic Stroke, TIA, Migraine or Decompression Illness
Acronym: Paradigm IV
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Cierra (Industry)
Responsible Party: Peggy McLaughlin, Cierra, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA0012
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: PFO; Stroke; Transient Ischemic Attack; Migraine; Decompression Illness
Keywords: PFO; Stroke; Transient Ischemic Attack; Migraine; Decompression Illness
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: PFx Closure System

SUMMARY:
The primary object of this study is to demonstrate the continued safety and performance of the PFx Closure System when utilized for patients with PFOs suffering from cryptogenic stroke, transient ischemic attack, migraine or decompression illness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years old
* PFO with one or more of:

  * Cryptogenic stroke,
  * TIA or embolism,
  * History of severe migraine headaches, or
  * History of severe decompression illness.

Exclusion Criteria:

* In appropriate anatomy (vascular or cardiac) or inappropriate medical condition for PFO closure and study medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-08; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
PFO closure at 6 months post procedure. | 6 months post procedure

SECONDARY OUTCOMES:
PFO closure at 30 days and 12 months post procedure. AE event rate for all subjects. Measurement of migraine severity or frequency at 6 and 12 months post procedure for subjects enrolled due to diagnosis of migraine. | 30 days; 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Horst Sievert, MD, Principal Investigator — Cardiovascular Center Frankfurt, Germany
Locations (1):
- Cardiovascular Center Frankfurt Sankt katharinen, Frankfurt, Germany